CLINICAL TRIAL: NCT03747562
Title: Multi-centre, Double-blind, Randomized-controlled Trial to Study the Efficacy and Safety of Gabapentin to Reduce Strong Opioid Use in Treatment of Radiation-induced Pain in Head and Neck Cancer Patients During Curative Radio(chemo)therapy.
Brief Title: Study of Efficacy and Safety of Gabapentin to Reduce the Need for Strong Opioid Use in Head and Neck Cancer Patients.
Acronym: stREnGTH
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University Hospital, Ghent (Other)
Collaborators: General Hospital Groeninge (Other); KU Leuven Campus Kulak Kortrijk (Unknown); Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-2657
Record Dates: First submitted 2018-10-09; First posted 2018-11-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Head Neck Cancer; Radiation Neuropathy; Pain, Neuropathic
Keywords: Gabapentin
MeSH Terms: conditions — Head and Neck Neoplasms; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Randomised-controlled trial where patients are randomised to either the experimental group (E) receiving gabapentin or the control group (C) receiving a matching placebo, both in addition to standard analgesic therapy (WHO ladder steps 2 and 3).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both patient groups will receive gabapentin or a matching placebo additional to the standard analgesic therapy, and will be asked to consume the content following the predefined directions provided to them. Both the investigators and the patients will be blinded for the IMP, since gabapentin and the matching placebo will appear identical.
  The clinical pharmacist responsible for clinical trials as well as Bimetra clinics will receive a sealed envelope from the statistician with the information necessary for decoding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients randomised to the experimental group will receive a prescription for a gabapentin starting dose of 100 mg three times a day (ter in die, t.i.d) /day per orally, additional to the analgesics according to standard local practices.
  Gabapentin dosage may be gradually increased based on individual patient response and tolerability, and as per standard practice in accordance with the drug label. The dose can be further increased in 300 mg/day increments (dose increments of 50% - 100%) every two to three days, up to a maximum dose of 3600 mg/day. The minimum time to reach a dose of 1800 mg/day is one week, to reach 2400 mg/day is a total of two weeks, and to reach 3600 mg/day is a total of three weeks.
  Interventions: Drug: Gabapentin
- Control group (Placebo Comparator): Patients randomised to the control group will receive a prescription for a matching placebo. The starting dose will be the same as in the experimental group (100 mg three times a day per orally), additional to the analgesics according to standard local practices. Placebo can optionally follow the same dose scheme as described in the experimental arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin will be administrated orally, with or without food, and should be swallowed with sufficient fluid intake (e.g. a glass of water). Since head and neck cancer patients frequently experience swallowing difficulties, gabapentin capsules will be provided to enable opening of the capsule and use of the contents for mixture with food or liquids. Moreover, gabapentin powder can be dissolved in water to enable injection of the drug into a percutaneous endoscopic gastrostomy tube.
  Arms: Experimental group
Other: Placebo — Placebo will be administrated orally, with or without food, and should be swallowed with sufficient fluid intake (e.g. a glass of water). Since head and neck cancer patients frequently experience swallowing difficulties, placebo capsules will be provided to enable opening of the capsule and use of the contents for mixture with food or liquids. Moreover, placebo powder can be dissolved in water to enable injection of the drug into a percutaneous endoscopic gastrostomy tube.
  Arms: Control group

SUMMARY:
A multi-centre, double-blind, randomized-controlled trial to study the efficacy and safety of gabapentin to reduce the need for strong opioid use in the treatment of radiation-induced pain in head and neck cancer (HNCA) patients undergoing a curative 7-week radio(chemo)therapy course with curative intent. The aim of this study is to establish if addition of gabapentin is more effective in reducing the need to start (or dosage-increase) a strong opioid for HNCA pain than a matching placebo additional to standard pain management (WHO-ladder step 2 and 3).

DETAILED DESCRIPTION:
Although pain is a major symptom in head and neck cancer (HNCA) patients, few studies focus on pain management in this population. Current optimal HNCA pain control usually requires the use of a strong opioid (WHO-ladder step 3), increasing the risk of opioid side effects and toxicities. Gabapentin, originally an anticonvulsant drug, has been effectively used off-label to treat multiple neuropathic pain syndromes such as cancer pain, and has been suggested to reduce the need for high doses of strong opioids in HNCA patients under radio(chemo)therapy. A multi-centre, phase III, double-blind, randomised-controlled trial will be set up randomising patients between the experimental group (E) receiving gabapentin, or the control group (C) receiving a matching placebo, both in addition to standard analgesic therapy (steps 2 and 3 on WHO-ladder). The investigators aim to establish if addition of gabapentin is more effective in reducing the need to start (or dosage-increase) a strong opioid for HNCA pain than a matching placebo additional to standard pain management (WHO-ladder step 2 and 3), in HNCA patients scheduled for a curative 7-week radio(chemo)therapy course.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck region, generally cancer of the oral cavity, pharynx and larynx. Cancer of the nasal cavity, nasopharynx, paranasal sinuses, parotid gland, or a T1-2N0M0 of the glottis are excluded.
* Primary cancer eligible for primary or adjuvant radiotherapy with or without systemic treatment, with curative intent
* TNM stage I to IVb, without distant metastases
* Patients should require the intake of at least a weak opioid (inclusion starting at prescription/intake of at least a step 2 drug (e.g. a step 2 or step 3 analgesic; if a physician would decide to skip step 2) according to the WHO pain ladder)
* Patients should be 18 or older at the time of enrolment
* Patients should be able to adequately communicate in Dutch or French

Exclusion Criteria:

* Patients younger than 18 years at the time of enrolment
* Patients with cancer of the nasal cavity, nasopharynx, paranasal sinuses, parotid glands, or a T1-2N0M0 of the glottis
* Pregnant or lactating women (Non-pregnancy must be confirmed before the first administration by use of a urine pregnancy test. Any positive urine pregnancy test must be confirmed via a serum β-HCG test).
* Patients presenting with another non-cured cancer (e.g. PSA or CEA not within normal range as determined by the treating physician)
* Patients with a prior history of cancer, with or without radio(chemo)therapy, diagnosed within the last 5 years
* Patients who report post-operative pain, as judged by the investigator
* Patients with a locoregional relapse of a prior head and neck tumour, for which they already received surgery or radio(chemo)therapy
* Patients who received radiation therapy in the head and neck region in the past
* Patients with (severe) dementia (DSM-IV criteria) or other significant psychiatric illnesses (e.g. mania, psychosis, schizophrenia, Korsakov, diagnosed major depression and/or history of suicide attempts) that would preclude study compliance
* Patients taking gabapentin/pregabalin or with prior gabapentin/pregabalin use
* Patients taking pain medications (e.g. topical analgesics such as lidocaine gel or lidocaine patch) for pre-existing pain of other aetiology. Administration of topical mouthwash is allowed.
* Patients with pre-existing peripheral neuropathy of another aetiology, B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning, syphilis, amyloidosis, hyper- or hypothyroidism, inherited neuropathy
* Patients taking anti-epileptics for (myoclonic) seizures or neuropathic pain
* Patients taking anti-depressants for neuropathic pain (i.e. anti-depressant described as the first and second group in the BCFI are excluded, anti-depressants of the third group or selective serotonin reuptake inhibitors (SSRI) are allowed)
* Patients with chronic kidney failure (creatinine clearance <30 ml/min)
* Patients with a diagnosis of acute pancreatitis within the last 6 months
* Patients with a current active hepatic or biliary disease
* Patients presenting with clinical signs of CNS depression
* Patients with a hypersensitivity to the active substance
* Patients with galactose intolerance and/or lactase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Requirement of patients included in 7-week curative radio(chemo)therapy for a (dose-escalation of) strong opioid | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Through pain diary, weekly visit by doctor and research assistant, the need for (dose-escalation of) strong opioid will be assessed.

SECONDARY OUTCOMES:
Pain prevalence, prevalence of opioid use within HNCA patients | Daily, weekly and assessed at visit 1 (moment of inclusion), visit 2 (anticipated week 5), visit 3 (end of radio(chemo)therapy), and week 24 (follow-up)
  Through pain diary, weekly visit by doctor and research assistant, patients will be asked to rate their pain
Maintenance or amelioration of pain within subtypes measured by the 0-10 numeric visual analogue pain rating scale. | Daily, weekly and assessed at visit 1 (moment of inclusion), visit 2 (anticipated week 5), visit 3 (end of radio(chemo)therapy), and week 24 (follow-up)
  Pain assessment of subtypes of patients, according to their tumour location, through the 0-10 numeric visual analogue pain rating scale. This scale is a tool to measure the pain of patients, with a score of 0 if the patient has no pain, a score of 5 if the patient has moderate pain and a score of 10 if the patient copes with the worst possible pain. So higher values represent worse pain.
Maintenance or amelioration of pain within subtypes measured by the Neuropathic Pain Scale | Daily, weekly and assessed at visit 1 (moment of inclusion), visit 2 (anticipated week 5), visit 3 (end of radio(chemo)therapy), and week 24 (follow-up)
  Pain assessment of subtypes of patients, according to their tumour location, through the Neuropathic Pain Scale. Patients give a score between 0 until 10 on different aspects of pain as pain sharpness, heat/cold, dullness, intensity, unpleasantness, and surface vs. deep pain which all represent the subtypes of the Neuropathic Pain Scale. A score between 0 and 10 will be assigned to these different subtypes of pain, with a score of 0 if the patient has no pain, a score of 5 if the patient has moderate pain and a score of 10 if the patient copes with the worst possible pain. So higher values represent worse pain. The scores on all these subscales are not combined as we are interested in the subtypes of pain themselves.
Maintenance or amelioration of pain within subtypes measured by the Brief Pain Inventory (Short Form). | Daily, weekly and assessed at visit 1 (moment of inclusion), visit 2 (anticipated week 5), visit 3 (end of radio(chemo)therapy), and week 24 (follow-up)
  Pain assessment of subtypes of patients, according to their tumour location, through the Brief Pain Inventory (Short Form).
Effect on treatment-related toxicity (mucositis, dysphagia, fatigue, weight loss) | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Treatment-related toxicities will be scored by the local physician
Effect on hospitalisation requirement | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Effect on hospitalisation will be assessed by the local physician and the research assistant
Effect on percutaneous endoscopic gastrostomy tube placement | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Effect on the placement of percutaneous endoscopic gastrostomy tube will be assessed by the local physician and research assistant
Difference in dose of opioids needed for pain relief between the experimental and control group | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Monitoring of opioid therapy until primary endpoint
Effect on quality of life, and sleep quality in specific, of head and neck cancer patients assessed by EORTC QLQ C30 | Visit 1 (moment of inclusion), visit 2 (anticipated week 5), visit 3 (end of radio(chemo)therapy), and week 24 (follow-up)
  Measured by EORTC QLQ C30
Effect on quality of life, and sleep quality in specific, of head and neck cancer patients assessed by HN35 Questionnaires | Visit 1 (moment of inclusion), visit 2 (anticipated week 5), visit 3 (end of radio(chemo)therapy), and week 24 (follow-up)
  Measured by HN35 Questionnaires
Effect on quality-adjusted life years | Visit 1 (moment of inclusion), visit 2 (anticipated week 5), visit 3 (end of radio(chemo)therapy), and week 24 (follow-up)
  Measured by EuroQoL
Drug tolerance | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Monitoring of drug tolerance by local physician on weekly visits. The effects of the drug can either be unchanged, lessened, or increased. According to this, the physician will adapt the dose for patient. This will be weekly reported by the local physician to the research associate.
(S)AE | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Monitoring of drug safety by local physician according to treatment-related toxicities, scored weekly by the local physicians according to the Common Terminology Criteria of Adverse Events (NCI CTCAE 5.0). Analgesic-induced side effects will be evaluated with regard to nausea, constipation, sleepiness, dizziness, confusion, hypersensitivities, urinary retention, pruritus and respiratory depression.
Acceptance rate of gabapentin | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Weekly monitoring of drug compliance by local physician and research associate. Research associate counts amount of medication (gelules) that are left to assure there is therapy compliance.
Ease of use of trial medication | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Through pain diary, weekly visit by research assistant, patients will be asked about the ease of use of trial medication
Study drop-out | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Continuous follow-up of patients (weekly or daily) by research assistant
Patient satisfaction | Continuous monitoring from patient enrollment until week 7 or date of requiring a (dose-escalation of) strong opioid if this occurs before week 7 (end of radio(chemo)therapy)
  Through weekly visit by research assistant, patients will be asked how satisfied they are with current trial medication
Selection of biomarkers to identify patients prone to develop HN cancer pain/treatment-related pain | At time of patient enrollment
  Patients will be able to agree or disagree with the collection of blood samples on the informed consent form as these translational aspects are not an obligatory part of this trial. In patients who give their consent, one SST blood sample and one EDTA blood sample will be collected at the time of inclusion.
Selection of biomarkers to select patients who benefit more from analgesic treatment with gabapentin | At time of patient enrollment
  Patients will be able to agree or disagree with the collection of blood samples on the informed consent form as these translational aspects are not an obligatory part of this trial. In patients who give their consent, one SST blood sample and one EDTA blood sample will be collected at the time of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Boterberg, MD, PhD, Principal Investigator — Head of Clinic, Radiation Oncologist Department of Radiation Oncology
Locations (2):
- Belgium (2):
  - UZ Ghent, Ghent, Oost-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: No